CLINICAL TRIAL: NCT00003702
Title: A Randomized Phase III Trial of Weekly Parenteral Methotrexate Versus "Pulsed" Dactinomycin as Primary Management for Low Risk Gestational Trophoblastic Neoplasia
Brief Title: Methotrexate Compared With Dactinomycin in Treating Patients With Gestational Trophoblastic Neoplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: Eastern Cooperative Oncology Group (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0174; NCI-2011-02026 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-G174; CDR0000066809; GOG-0174 (Other: Gynecologic Oncology Group); GOG-0174 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2018-05-15 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2016-02

CONDITIONS: Good Prognosis Metastatic Gestational Trophoblastic Tumor; Hydatidiform Mole; Non-Metastatic Gestational Trophoblastic Tumor; Uterine Corpus Choriocarcinoma
MeSH Terms: conditions — Hydatidiform Mole | interventions — Dactinomycin; Methotrexate; merphos

ARMS (2):
- Arm I (methotrexate) (Experimental): Patients receive methotrexate intramuscularly once weekly in the absence of disease progression or unacceptable toxicity. Patients continue on treatment until 1 beta HCG titer is below the institutional normal. Patients then receive 1 additional consolidation treatment.
  Interventions: Drug: Methotrexate
- Arm II (dactinomycin) (Experimental): Patients receive dactinomycin IV over 15 minutes every 2 weeks in the absence of disease progression or unacceptable toxicity. Patients continue on treatment until 1 beta HCG titer is below the institutional normal. Patients then receive 1 additional consolidation treatment.
  Interventions: Biological: Dactinomycin

INTERVENTIONS:
Biological: Dactinomycin — Given IV
  Other Names: Actinomycin A IV; Actinomycin C1; ACTINOMYCIN D; Actinomycin I1; Actinomycin IV; Actinomycin X 1; Actinomycin-[thr-val-pro-sar-meval]; Cosmegen; DACT; Dactinomycine; Lyovac Cosmegen; Meractinomycin
  Arms: Arm II (dactinomycin)
Drug: Methotrexate — Given intramuscularly
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
  Arms: Arm I (methotrexate)

SUMMARY:
Randomized phase III trial to compare the effectiveness of methotrexate with that of dactinomycin in treating patients who have gestational trophoblastic neoplasia. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether methotrexate is more effective than dactinomycin in treating patients with gestational trophoblastic neoplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare the efficacy of methotrexate vs dactinomycin, as measured by complete response rate, in patients with low-risk gestational trophoblastic neoplasia.

II. Compare the toxicity of these regimens in these patients. III. Determine whether the definition of persistent gestational trophoblastic neoplasia is accurate (as determined by the likelihood that the beta human chorionic gonadotropin [HCG] titer would decline on the day treatment is initiated).

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive methotrexate intramuscularly once weekly in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive dactinomycin IV over 15 minutes every 2 weeks in the absence of disease progression or unacceptable toxicity. All patients continue on treatment until 1 beta human chorionic gonadotropin (HCG) titer is below the institutional normal. Patients then receive 1 additional consolidation treatment.

Patients are followed every 4 weeks for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven low-risk gestational trophoblastic neoplasia (persistent hydatidiform mole or choriocarcinoma), defined as 1 of the following:

  * Less than 10% decrease in the beta human chorionic gonadotropin (HCG) titer over 3 weekly titers
  * Greater than 20% sustained rise in beta HCG titer over two consecutive weeks
  * Persistently elevated beta HCG titer more than 4 months after initial curettage (greater than 5 mIU/mL minimum)
  * Histologically proven nonmetastatic choriocarcinoma
  * Metastases to vagina, parametria, or lung (if no single pulmonary lesion is greater than 2 cm)
* WHO score 0-6 (not including blood group or CT lung)
* No histologically confirmed placental site pseudotumor
* Must have undergone at least 1 uterine curettage
* Previously untreated disease
* Performance status - GOG 0-2
* WBC at least 3,000/mm^3
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGPT and SGOT no greater than 3 times ULN
* Alkaline phosphatase no greater than 3 times ULN
* No significant prior abnormal hepatic function
* Creatinine no greater than 2.0 mg/dL
* No significant prior abnormal renal function
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for one year after study entry
* No other prior or concurrent malignancies within the past 5 years except nonmelanomatous skin cancer
* No prior chemotherapy for gestational trophoblastic neoplasia
* No concurrent curettage except as needed to control vaginal bleeding or to rule out placental site pseudotumor

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 1999-06; Primary Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Osborne, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial opened to patient accrual on 6/14/1999 and closed to accrual on 2/26/2007.
Groups:
- Arm 1: Methotrexate 30 mg/m2 IM Weekly: Arm 1: Methotrexate 30 mg/m2 IM weekly
- Arm 2: Dactinomycin 1.25 mg/m2 IV Push Every 2 Weeks: Arm 2: Dactinomycin 1.25 mg/m2 IV push every 2 weeks
Period: Overall Study
Arm/Group | Arm 1: Methotrexate 30 mg/m2 IM Weekly | Arm 2: Dactinomycin 1.25 mg/m2 IV Push Every 2 Weeks
Started | 120 | 120
Completed | 107 | 109
Not Completed | 13 | 11
Not completed — Ineligible cell types | 2 | 2
Not completed — Did not meet criteria for persistence | 8 | 5
Not completed — WHO score > 6 | 2 | 1
Not completed — Inadequate documentation of disease | 1 | 3

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Methotrexate 30 mg/m2 IM Weekly | Arm 2: Dactinomycin 1.25 mg/m2 IV Push Every 2 Weeks | Total
Number analyzed (Participants) | 107 | 109 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (7.9) | 30.4 (8.6) | 29.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 109 | 216
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Based on Blood Human Chorionic Gonadotropin (hCG) Assay
Description: Primary outcome is measured as a difference in proportion responding between treatment arms and evaluated using a chi square test. A complete response was defined as a normal hCG sustained over four weekly measurements.
Time Frame: Endpoint was assessed by hCG measurements taken weekly, once normal, treatment was bi-weekly, then monthly, up to 12 months.
Population: Eligible patients who received a random treatment allocation
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Methotrexate 30 mg/m2 IM Weekly | Arm 2: Dactinomycin 1.25 mg/m2 IV Push Every 2 Weeks
Number analyzed (Participants) | 107 | 109
Participants
  Complete/Cure | 57 | 76
  Non-response | 48 | 29
  Inevaluable | 2 | 4

2. Primary Outcome: Incidence of Adverse Effects (Grade 3 or Higher) as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 2.0
Description: Number of participants with a maximum grade of 3 or higher during the treatment period.
Time Frame: Prior to study entry, weekly during treatment, up to 12 months after normal titer, an average of 7 months.
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Methotrexate 30 mg/m2 IM Weekly | Arm 2: Dactinomycin 1.25 mg/m2 IV Push Every 2 Weeks
Number analyzed (Participants) | 107 | 109
Participants | 14 | 20

3. Secondary Outcome: Number of Patients With a Decline of hCG on Day 1 of Treatment
Description: Number of patients with a decline in hCG on day 1 of treatment relative to the level at enrollment. A decline is defined as a decrease by 1 or more units between enrollment and treatment start.
Time Frame: Prior to study entry and on Day 1 of treatment
Population: Eligible and evaluated patients
Measure: Count of Participants; unit: Participants
Groups:
- Enrolled Participants: Enrolled participants that had a subsequent hCG measurement after enrollment and before treatment
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 178
Participants | 72

ADVERSE EVENTS:
Time Frame: Through Study completion, an average of 7 months.
Description: The frequencies of any serious adverse event or other adverse events (grade 2 or higher) by category or specific term occurring during treatment and up to 30 days after stopping the study treatment are reported. Adverse events were collected by Organ System Class.
Arm/Group | Arm 1: Methotrexate 30 mg/m2 IM Weekly | Arm 2: Dactinomycin 1.25 mg/m2 IV Push Every 2 Weeks
Serious Adverse Events (participants affected / at risk) | 0/107 | 1/107
Other Adverse Events (participants affected / at risk) | 50/107 | 68/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Methotrexate 30 mg/m2 IM Weekly (N=107) | Arm 2: Dactinomycin 1.25 mg/m2 IV Push Every 2 Weeks (N=107)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Methotrexate 30 mg/m2 IM Weekly (N=107) | Arm 2: Dactinomycin 1.25 mg/m2 IV Push Every 2 Weeks (N=107)
Leukopenia (Blood and lymphatic system disorders) | 3 | 7
Neutropenia (Blood and lymphatic system disorders) | 6 | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Anemia (Blood and lymphatic system disorders) | 7 | 14
Other Hemotologic (Blood and lymphatic system disorders) | 0 | 1
Allergy (Immune system disorders) | 2 | 0
Auditory (Ear and labyrinth disorders) | 1 | 1
Cardiovascular (Cardiac disorders) | 0 | 2
Coagulation (Vascular disorders) | 1 | 0
Constitutional (General disorders) | 12 | 15
Dermatologic (Skin and subcutaneous tissue disorders) | 1 | 0
Endocrine (Endocrine disorders) | 0 | 2
Gastrointestinal (Gastrointestinal disorders) | 7 | 14
Nausea (Gastrointestinal disorders) | 8 | 21
Vomiting (Gastrointestinal disorders) | 3 | 14
Diarrhea (Gastrointestinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 5 | 1
Genitourinary/Renal (Renal and urinary disorders) | 3 | 0
Hemorrhage (Blood and lymphatic system disorders) | 9 | 13
Hepatic (Hepatobiliary disorders) | 2 | 3
Infection/Fever (Infections and infestations) | 7 | 4
Metabolic (Metabolism and nutrition disorders) | 0 | 2
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 | 0
Neurologic (Nervous system disorders) | 6 | 5
Ocular/Visual (Eye disorders) | 5 | 4
Pain (General disorders) | 13 | 14
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 | 8
Sexual (Reproductive system and breast disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less